CLINICAL TRIAL: NCT01041677
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-Center Study to Evaluate the Effect of JNJ-16269110 on Hepatic Triglyceride Content in Obese Subjects
Brief Title: A Study of the Safety of R256918 in Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013735
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Nutritional and Metabolic Diseases; Metabolic Diseases; Nutrition Disorders; Overweight
Keywords: Obesity; Overweight; Body Weight; Body Size; Nutritional and Metabolic Diseases
MeSH Terms: conditions — Obesity; Nutritional and Metabolic Diseases; Metabolic Diseases; Nutrition Disorders; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 001 (Experimental): R256918 10 mg capsule twice daily
  Interventions: Drug: R256918
- 002 (Experimental): R256918 15 mg capsule twice daily
  Interventions: Drug: R256918
- 003 (Placebo Comparator): placebo placebo capsule twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: R256918 — 10 mg capsule twice daily
  Arms: 001
Drug: placebo — placebo capsule twice daily
  Arms: 003
Drug: R256918 — 15 mg capsule twice daily
  Arms: 002

SUMMARY:
This study investigates the safety of 12 weeks of treatment with R256918, in obese patients (JNJ-16269110 and R256918 are different names for the same molecule). The primary objective of the study is to investigate mean changes in Hepatic Triglyceride Content (HTGC), which is the fat content of the liver, from baseline to week 6 and 12 by 1H-Magnetic Resonance Spectroscopy (MRS), a specialized non invasive radiology test. Additional measures include body mass index (BMI), fasting glucose,lipid levels, and blood pressure. Safety assessments performed during the trial include laboratory tests, vital sign measurements, and adverse event reporting.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither physician nor patient knows the name of the assigned drug), placebo-controlled , parallel-group study with 3 treatment arms, each consisting of 27 obese patients. The study will include 3 phases - pretreatment, double-blind and posttreatment . During the pretreatment phase patients undergo general screening assessments and if eligible, Magnetic Resonance Spectroscopy (MRS) screening will be performed. During the double-blind treatment phase patients will receive dietary counseling, study medication, have urine and blood laboratory tests, a follow up MRS examination and have regular clinic visits for symptoms assessment. The double blind treatment phase ends with an end-of-treatment or early withdrawal visit. A patient withdrawing from the study prior to the end of the 12 week treatment phase will attend an early withdrawal visit, which is the same as the end-of-treatment visit. This visit will include laboratory tests and a follow up MRS examination. Post-treatment: A follow-up evaluation will occur 14 days after the end of treatment. Study visits are scheduled to occur nearly every 14 days following the baseline visit in week 1. The total study duration is approximately 15 weeks. The study will include the following evaluations of safety and tolerability: mean percent change in liver fat content at week 6 and week 12 or at the end of the patients participation in the study, in case of early withdrawal. Safety evaluations for the study will include the monitoring of adverse events, clinical laboratory tests including pregnancy testing, electrocardiograms (ECGs), vital sign measurements (pulse and blood pressure), physical examination, and patient reported assessment of GI symptoms. Special clinical laboratory safety tests will assess blood clotting or coagulation status, essential fatty acid status, lipid-soluble vitamin status: vitamin A, vitamin D, vitamin E, vitamin K, vitamin A/total cholesterol ratio, vitamin E/total cholesterol ratio and liver function tests. 10 mg capsules, 15 mg capsules, or matching placebo capsules taken orally.

ELIGIBILITY:
Inclusion Criteria:

* Liver fat content (HTGC) between 3% and 15%
* Obese defined as BMI between 30 and 50 kg/square meter
* Fasting plasma glucose < 7.0 mmol/liter

Exclusion Criteria:

* History of Obesity with a known cause (eg. Cushings disease)
* Diabetes Mellitus
* Weight reducing diet or receiving drugs to treat obesity within 3 months prior to screening
* Significant change in smoking habits within 3 months before enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Hepatic Triglyceride Content (HTGC) as measured by 1H-Magnetic Resonance Spectroscopy (MRS). | Baseline, 6 weeks, 12 weeks

SECONDARY OUTCOMES:
Change in Body weight | Baseline, weeks 1, 2, 4, 6, 8,10,12,14
Change in alanine aminotransferase and aspartate aminotransferase | Baseline, weeks 4, 6, 8,12,14
Changes in fasting glucose and insulin | Baseline, weeks 6, 12
Changes in systolic and diastolic blood pressure | Baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14
Changes in total-, HDL- and LDL-cholesterol and triglycerides | Baseline, weeks 6,12

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (3):
- Helsinki, Finland
- Zuidlaren, Netherlands
- Gothenburg, Sweden

REFERENCES:
- See also: A Study of the Safety of R256918 in Obese Patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=762&filename=CR013735_CSR.pdf